CLINICAL TRIAL: NCT01187888
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Assess the Efficacy, Safety and Tolerability of Rasagiline in Subjects With Progressive Supranuclear Palsy (Phase III)
Brief Title: Efficacy, Tolerability and Safety of Azilect in Subjects With Progressive Supranuclear Palsy
Acronym: PROSPERA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: IMP used off label by phys. in pat. with PSP. Thus no more eligible patients were available for the study(pre-treatm.with Rasagiline=exclusion criterion
Sponsor: Prof. Dr. Stefan Lorenzl (Other)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Stefan Lorenzl, Principal Investigator and Sponsor Delegated Person, Hospital of the University of Munich, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08P02; 2008-007520-26 (EudraCT Number)
Record Dates: First submitted 2010-08-20; First posted 2010-08-24 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Progressive Supranuclear Palsy
Keywords: PSP; Progressive Supranuclear Palsy; Rasagiline; Azilect; PROSPERA
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — rasagiline; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rasagiline (Active Comparator)
  Interventions: Drug: Rasagiline
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Rasagiline — tablet once daily 1 mg 1 year
  Other Names: Azilect
  Arms: Rasagiline
Drug: Sugar pill — tablet once daily one year
  Other Names: Placebo
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to determine whether rasagiline is effective in the treatment of Progressive Supranuclear Palsy (PSP), a rapidly progressing disease with a symptomatology similar to Parkinson's Disease. The major aim of this study is the limitation or halting of the process of neurodegeneration and influence postural instability.

DETAILED DESCRIPTION:
Progressive Supranuclear Palsy (PSP) is a rapidly progressing disease with a median survival after onset of symptoms of 5.8 years.PSP is characterized by early falls, vertical ophthalmoparesis, akinetic-rigid features, prominent bulbar dysfunction and fronto-subcortical dementia. So far there is no treatment for the disease as the negative outcomes of the vast majority of studies make it impossible to set standards. As the majority of patients experience severe falls and vertigo already in the early phase of the disease, the drug of desire would be able to slow disease progression with a special focus on postural instability and exert neuroprotective effects. The monoamino oxidase inhibitor Rasagiline might be able to influence progression of PSP.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs of Progressive Supranuclear Palsy (PSP). Diagnosis will be made for patients with clinical probable PSP (Litvan et al., 1996). Patients will be included with PSP stage </= II (Golbe et al., 1997), at least with a PSPRS < 40 (Golbe et al., 2007) and according to the diagnostic criteria resumed after the Neuroprotection and Natural History in Parkinson Plus Syndromes (NNIPPS) trial (Bensimon et al., 2009)
* Patients, male or female, aged 50 to 80 years
* Subjects whose clinical condition at the time of enrolment does not or requires a low [</= 500 mg /day] stable dose of L-3,4-Dihydroxyphenylalanine (L-DOPA) for at least 2 weeks prior to study entry
* Capability and willingness to give written signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study

Exclusion Criteria:

* No clinically probable PSP
* No written informed consent possible
* Age > 80 or < 50 years
* Dementia (Mini-Mental State Examination [MMSE] </= 24)
* Subjects with clinically significant psychiatric illness, including major depression
* Subjects who have taken any experimental drugs within 60 days prior to baseline
* Subjects who have used sympathomimetics (including over-the-counter remedies - nasal or oral), dextromethorphan, pethidine or St. John's wort within 7 days prior to baseline.
* Loss of postural reflexes (no independent walking possible, inability to stand unassisted, wheelchair-bound)
* Feeding tube / recommendation for a feeding tube
* Unintelligible speech
* History of brain disease (e.g. repeated strokes, cerebral tumour, hydrocephalus)
* 1-methyl-4-phenyl-1,2,5,6-tetrahydropyridine (MPTP) exposure
* Oculogyric crisis
* Early severe autonomic failure
* Systemic disorder affecting the brain
* Women who are not postmenopausal (e.g. one year without menstrual periods) or surgically sterilized.
* Known history of hypersensitivity to the investigational drug or to drugs with a similar chemical structure
* Subjects who have used antidepressants, including selective serotonin re-uptake inhibitors, tricyclic and tetracyclic antidepressants (except amitriptyline <= 50 mg/day, trazodone < = 100 mg/day, citalopram < = 20 mg/ day, sertraline < = 100 mg/day and paroxetine < = 30 mg/day, escitalopram < = 10 mg/day) within 42 days prior to baseline
* Subjects who have used any drugs known to have been involved in a drug interaction via inhibition of hepatic Cytochrome P450 1A2 (CYP 1A2) within 30 days prior to baseline (cimetidine, ciprofloxacin, clarithromycin, enoxacin, erythromycin, fluvoxamine, isoniazide, nalidixic acid, norfloxacin, troleandomycin, zileuton)
* Subjects who have used Monoamine oxidase (MAO) inhibitors including reserpine and methyldopa within three months prior to baseline
* Anti-emetic or antipsychotic medication with central dopamine antagonist activity (except quetiapine fumarate) within six months prior to baseline
* Participation in a clinical trial within the last 30 days prior to study start
* Unstable antiparkinsonian medication within 30 days before baseline
* Previous use of Rasagiline or Selegiline
* Subjects who have a clinically significant or unstable medical or surgical condition that may preclude safe and complete study participation (based on the investigator's judgment). Such conditions might include cardiovascular, vascular diseases, pulmonary, hepatic impairment (Child-Pugh score > 5), renal, or metabolic dis-eases or malignancies as determined by medical history, physical examination, laboratory tests, or ECG

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Assessment of the need for additional L-DOPA therapy or the need to increase the dose of L-DOPA during the trial | 1 year
  Since there is no established treatment regimen for Progressive Supranuclear Palsy (PSP) patients, the only well characterized medication is L-3,4-Dihydroxyphenylalanine (L-DOPA) therapy. Since this therapy may exert a small effect in PSP patients, begin with L-DOPA therapy or increase in L-DOPA therapy will be used in this trial as rescue medication.
Reduction of the reported deterioration using the PSP rating scale | 1 year
  To assess the efficacy of Rasagiline using the Progressive Supranuclear Palsy Rating Scale (PSPRS), aiming at a 33% reduction of the reported deterioration (Golbe et. al., 2007), i.e. a mean yearly increase of 6.5 instead of 9.7 points.

SECONDARY OUTCOMES:
Reduction of gait disturbances and postural stability | 1 year
Adverse Event (AE) incidence | 1 year
Safety laboratory values (blood cell count, aspartate aminotransferase [AST], alanine aminotransferase [ALT], creatinine, Vitamin B12, folic acid, homocysteine and methylmalonic acid) | 1 year
Vital signs | 1 year
Number of subjects (%) who discontinue the study | 1 year
Number of subjects (%) who discontinue the study due to AEs | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Lorenzl, PD Dr., Principal Investigator — Klinikum der Universität München (Hospital of the University of Munich)
Locations (1):
- Department of Neurology and Palliative Care Klinikum der Universität München (Hospital of the University of Munich), München, Germany